CLINICAL TRIAL: NCT06414018
Title: Effect of Equivalent Dose of Alfentanil and Sufentanil Combined With Remimazolam in Complex Bronchoscopic Treatment
Brief Title: Effect of Equivalent Dose of Alfentanil and Sufentanil in Bronchoscopic Treatment
Acronym: EOEDSAAIBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Xinxiang Central Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, clincal doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EEDSA
Record Dates: First submitted 2024-05-10; First posted 2024-05-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Effect of Drug
Keywords: Afentanil; sufentanil; bronchoscopy; Recovery time
MeSH Terms: interventions — Alfentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil group (Experimental): The dose of sufentanil group is 0.2μg/kg
  Interventions: Drug: Alfentanil
- Alfentanil (Experimental): The dose of aifentanil group is 10μg/kg
  Interventions: Drug: Alfentanil

INTERVENTIONS:
Drug: Alfentanil — alfentanil 10ug/kg is used for anesthesia induction
  Other Names: sufentanil

SUMMARY:
The equivalent dose of sufentanil and afentanil combined with laryngeal mask was used for complex bronchoscopy to observe the intraoperative effect and the influence on the recovery of patients

DETAILED DESCRIPTION:
Afentanil is a powerful, fast-acting narcotic analgesic, which can effectively inhibit intubation reflex. Compared with sufentanil, it has a short half-life and is safer, and can be used as the first choice for short surgical analgesics. In this study, by comparing the use of equivalent dose sufentanil and afentanil combined with laryngeal mask for complex bronchoscopy, the intraoperative analgesic effect and the influence on the recovery of patients were observed, and a better anesthesia scheme was provided for tracheoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80,
* ASA I-III level;
* BMI 18.5~23.9;

Exclusion Criteria:

* Patients with full stomach and high risk of reflux aspiration;
* Allergic to benzodiazepines, opioids, rocuronium bromide;
* Those who have taken sedative, analgesic or antidepressant drugs within 24 hours;
* Pregnant and lactating women;
* severe liver and kidney dysfunction;
* Patients with severe anemia and hypoproteinemia;
* Previous drug use history;
* Recently participated in other clinical studies;
* Patients who cannot cooperate with communication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
time of Recovery | 1day
  the time from the end of surgery to awake of patient

SECONDARY OUTCOMES:
Time records | 1 day
  Anesthesia time, induction time, surgical time, awakening time and recovery time
dose of drugs | 1 day
  The total amount of sedative and analgesic drugs used.
rate of respiratory suppression incidence | 1 day
  Respiratory frequency<8 times/min or SP02<90%
rate of Incidence of Treatment-Emergent Adverse Events | 1day
  Intraoperative blood pressure and heart rate changes: record the patient's intraoperative blood pressure, heart rate, and the use of related vasoactive drugs; Postoperative adverse reactions: such as hypertension, hypotension, tachycardia, gastrointestinal symptoms, postoperative restlessness, etc

OTHER OUTCOMES:
rate of Postoperative adverse reaction | 1 day
  Airway obstruction, hypoxemia, apnea, laryngeal spasm, bronchospasm, cough, postoperative nausea and vomiting, postoperative pain (VAS score), hypotension, bradycardia, dizziness

CONTACTS AND LOCATIONS:
Overall Officials: aijun xu, Dr, Principal Investigator — Tongji Hospital
Locations (1):
- Aijun Xu, Hubei, Wuhan, China

IPD SHARING:
Plan to Share IPD: No
You can request it from the main researcher.